CLINICAL TRIAL: NCT05312723
Title: Sleep Disturbance in Chronic Rhinitis: Evaluation of Nasal Symptoms, Sleep Disorder Questionnaires, and Sleep Architecture in Allergic & Non-Allergic Rhinitis in Dr. Cipto Mangunkusumo Hospital
Brief Title: Sleep Disturbance in Chronic Rhinitis
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Nina Irawati, Head of Allergy Immunology Division, Otorhinolaryngology Head and Neck Surgery Department, Indonesia University
Other Study IDs: 20-01-0074
Record Dates: First submitted 2022-03-28; First posted 2022-04-05 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Sleep Disturbance
Keywords: allergic; nasal congestion; daytime sleepiness; polysomnography
MeSH Terms: conditions — Parasomnias; Nasal Obstruction; Disorders of Excessive Somnolence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rhinitis allergy: Patients with rhinitis symptoms and positive skin pric test to one or more allergens.
- Non-rhinitis allergy: Patients with rhinitis symptoms and negative skin pric test to one or more allergens.

SUMMARY:
The aim of this study is to evaluate the characteristic of sleep disturbance in allergic and non-allergic rhinitis in Dr. Cipto Mangunkusumo Hospital, Jakarta. A cross sectional analytic descriptive study with consecutive sampling was performed. A total of 22 chronic rhinitis patients, consisted of 11 allergic and 11 non-allergic rhinitis were evaluated of their sleep disturbance's characteristics.

DETAILED DESCRIPTION:
At first, all recruited subjects were evaluated for total nasal symptom scores (TNSS) and nasal obstruction symptoms evaluation scores (NOSE). Sleep disorder was assessed using Epworth Sleepiness Scale (ESS), Pittsburg Sleep Quality Index (PSQI) questionnaires, and polysomnography (PSG). Both the allergic and non-allergic rhinitis groups will be compared in terms of their sleep disturbance characteristics (from comparing ESS, PSQI, and PSG results).

ELIGIBILITY:
Inclusion Criteria:

* All male and female between 18-60 years old with chronic rhinitis symptoms and sleep disorder
* Did not receive intranasal steroid within the last one month
* Have psychiatric disorder

Exclusion Criteria:

* Polyp
* Nasal or sinonasal tumor
* Septum deviation
* Chronic rhinosinusitis
* Adenoid hypertrophy
* Tonsil hypertrophy
* Macroglossia
* Oropharyngeal tumor

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Allergic and non-allergic rhinitis patients
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Mean value of TNSS based on VAS symptoms | Evaluation is done at Day 1(cross-sectional)
  Clinical symptoms was evaluated by visual analogue scale (VAS) based on total nasal symptoms score (TNSS). Total nasal symptoms score are based on four symptoms, which are rhinorrea, sneezing, itchy nose, and nose obstruction. Each symptom will be given a score between 1 (most mild symptom) until 5 (most severe symptom). The minum score for VAS based on TNSS is 4 (most mild symptom) and the maximum score is 40 (most severe symptom). VAS score less than five indicates a controlled rhinitis symptoms, while ≥ 5 indicates that symptoms are not controlled.
Nasal obstruction symtpms evaluation (NOSE) score | Evaluation is done at Day 1 (cross-sectional)
  Nasal obstruction symptoms was evaluated by NOSE score. It evaluates 5 items that indicates nasal obstruction symptoms that was experienced in the past 1 month. Each item has a score range from 0 to 20. It has a minimum score of 0 and a maximum score of 100. Score 5-25 indicates mild nasal obstruction, score 30-50 indicates moderate nasal obstruction, score 55-75 indicates severe nasal obstruction, and score > 80 indicates extreme nasal obstruction.
Sleep quality from Epworth sleepiness scale (ESS) | Evaluation is done at Day 1 (cross-sectional)
  Sleep quality assessed by Epworth sleepiness scale. ESS is a self-administered questionnaire consisted of 8 questions. It assessed the chances of falling asleep while engaged in different activities. Each item scored 0-3, with a minimum score of 0 (low normal daytime sleepiness) and a maximum score of 24 (severe daytime sleepiness). In this study, the cut off is score 5-9 indicates mild daytime sleepiness and score > 10 indicates severe daytime sleepiness.
Sleep quality from Pittsburg Sleep Quality Index (PSQI) | Evaluation is done at Day 1 (cross-sectional)
  Sleep quality assessed by Pittsburg Sleep Quality Index. PSQI consisted of 10 questions. These 10 questions were divided to 7 components, including subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbance, use of sleep medication, and daytime dysfunction. Each component score range from 0-23. Total score can range from 0 to 21. Score < 5 indicates good sleep quality and > 5 indicates poor sleep quality
Objective sleep measurement using polysomnography (PSG) | Evaluation is done at Day 1 (cross-sectional)
  Sleep parameters were objectively measured using polysomnography (PSG). Sleep architecture was assessed using non-rapid eye movement (NREM)/ rapid eye movement (REM) and respiratory analysis was assessed using respiratory disturbance index - rapid eye movement (RDI-REM) and respiratory effort related arousals (RERA). All the parameters will be presented as numeric data.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Irawati, Principal Investigator — Indonesia University
Locations (1):
- RSUPN Dr. Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia